CLINICAL TRIAL: NCT00301431
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Adaptive Design, Efficacy and Tolerability Study of 4 Fixed Doses of DVS-233 in Adult Outpatients With Fibromyalgia Syndrome
Brief Title: Study Evaluating the Efficacy of DVS-233 in Fibromyalgia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A4-327
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Adults; Outpatients; Adult; Double-Blind Method
MeSH Terms: conditions — Fibromyalgia

INTERVENTIONS:
Drug: DVS-233

SUMMARY:
The purpose of this study is to determine if DVS-233 is safe and effective in the treatment of pain and other symptoms of fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia according to 1990 American College of Rheumatology (ACR) criteria

Exclusion Criteria:

* Other painful conditions that may make results difficult to interpret.
* Treatment with other drugs for fibromyalgia with 14 days of study start or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050
Dates: Start 2006-08; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in the daily pain score from baseline to study day 105 of therapy.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire and the Patient Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (55):
- United States (55):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Anaheim, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Walnut Creek, California
  - Denver, Colorado
  - Cromwell, Connecticut
  - Brooksville, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Palm Beach Gardens, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Rockville, Maryland
  - Boston, Massachusetts
  - Newton, Massachusetts
  - Lansing, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Clementon, New Jersey
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Harleysville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sellersville, Pennsylvania
  - West Reading, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Summerville, South Carolina
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Middleton, Wisconsin